CLINICAL TRIAL: NCT03954275
Title: Detailed Assessment of Augmented Renal Clearance in a Large Mixed Intensive Care Unit Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Hospital, Ghent (Other); University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Matthias Gijsen, Principal investigator, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S61364
Record Dates: First submitted 2019-05-03; First posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Critical Illness; Augmented Renal Clearance
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients with a CrCl24h: Patients admitted to any intensive care unit (surgical, medical or cardiac) and having at least one 24h creatinine clearance measurement available.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This multi-center retrospective cohort study presents a detailed assessment of augmented renal clearance (ARC) in a mixed population of adult critically ill patients. Epidemiology of ARC will be studied in detail in a very heterogeneous population. Risk factors for ARC will be identified and a predictive scoring system for ARC ready to use in clinical practice will be constructed and validated. Performance of estimators of kidney function will be measured and a cutoff for ARC will be determined for the best estimator. Finally clinical impact of ARC will be explored using vancomycine and aminoglycosides levels as surrogate marker.

DETAILED DESCRIPTION:
Augmented renal clearance will be assessed in detail in a very large and heterogeneous adult critically ill population. Analysis will be conducted retrospectively on a multi-center database collected by the M@tric research group. M@tric collects data from all intensive care units (surgical, medical, cardiac) in 3 Belgian University Hospitals (Leuven, Ghent, Antwerp).

Anonymised admission, demographic, clinical and laboratory data collected from 2013 until the present will be retrieved from the M@tric database. These data will then be coded and analysed in R statistical software. ARC will be defined based on a 24h creatinine clearance (CrCl24h) >=130ml/min/1.73m².

Epidemiology and risk factors for ARC will be studied in order to confirm and clarify past studies which have mostly been done in rather small and specific subsets of patients. A predictive algorithm for ARC will be trained and subsequently validated for use in clinical practice. Moreover this algorithm will be compared to existing scoring systems, which have not yet found their way into clinical practice. This algorithm will provide the ability to anticipate ARC on the intensive care unit. Also use of formulae estimating renal function will be evaluated in this population. These estimators will be compared to the CrCl24h, which is considered the golden standard in clinical practice. A cutoff for the best estimating formula in order to detect ARC will be calculated. Finally the impact of ARC on serum levels of hydrophilic molecules likes vancomycine and aminoglycosides will be studied. As this research follows a retrospective design these levels will be used a surrogate marker for clinical impact. This will potentially point out some opportunities for future research on the clinical impact of ARC.

ELIGIBILITY:
Inclusion Criteria:

* Having at least one 24h creatinine clearance measurement available

Exclusion Criteria:

* Any form of renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted at any intensive care unit (surgical, medical, cardiac) from the 3 participating centra (Leuven University Hospitals, Ghent University Hospital, Antwerp University Hospital) between 2013 and present
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
ARC incidence per day | Retrospective analysis between January 2013 and December 2015
  Incidence of ARC per 100 ICU days
ARC incidence per admission | Retrospective analysis between January 2013 and December 2015
  Incidence of ARC in % of ICU admissions: with ARC incidence defined as at least once, min. 50% of the measurements, 100% of the measurements during ICU admission)
Duration and course of ARC episodes | Retrospective analysis between January 2013 and December 2015
  ARC episodes: number of episodes (count), length of the episodes (days) and both combined to obtain relative contribution to ARC as a % ((count*length)/total ARC days)
ARC daily prevalence | Retrospective analysis between January 2013 and December 2015
  Daily prevalence of ARC (% of ARC days per ICU admission day)
Logistic regression with ARC as dependent variable | Retrospective analysis between January 2013 and December 2015
  Risk factors associated with ARC will be identified through logistic regression analysis on demographic and clinical data.
Predictive algorithm for ARC | Retrospective analysis between January 2013 and December 2015
  An algorithm predicting ARC on the next day(s) will be created using a backward selection logistic regression model on the risk factors associated with ARC detected in this study and/or in previously published studies.
Most precise formula using Bland-Altman agreement analysis | Retrospective analysis between January 2013 and December 2015
  Bland-Altman agreement analysis between CrCl24h and 3 commonly used serum creatinine based formulae estimating renal function (CKD-EPI, C&G, MDRD) will be used to identify the formula with the best precision (SD of the bias).
Performance of the best cutoff for ARC using ROC curve analysis | Retrospective analysis between January 2013 and December 2015
  Performance of the best cutoff for ARC using ROC curve analysis on the most precise formula estimating renal function.
Exploration of clinical impact of ARC via surrogate markers | Retrospective analysis between January 2013 and December 2015
  Vancomycin and aminoglycoside (amikacin & gentamycin) serum concentrations will be used as surrogate markers to evaluate potential clinical impact of ARC.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Spriet, PhD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
To be discussed

REFERENCES:
- [Derived] Gijsen M, Huang CY, Flechet M, Van Daele R, Declercq P, Debaveye Y, Meersseman P, Meyfroidt G, Wauters J, Spriet I. Development and External Validation of an Online Clinical Prediction Model for Augmented Renal Clearance in Adult Mixed Critically Ill Patients: The Augmented Renal Clearance Predictor. Crit Care Med. 2020 Dec;48(12):e1260-e1268. doi: 10.1097/CCM.0000000000004667. PMID 33048900